CLINICAL TRIAL: NCT01585298
Title: A 1-week, Open-label, Multi-center Study to Explore Conduction Abnormalities During First Dose Administration of Fingolimod in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: STudy to vAlidate telemetRic ECG Systems for firsT Dose Administration of Fingolimod (START)
Acronym: START
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DDE17
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Fingolimod; Gilenya; ECG; Bradyarrythmia; conduction abnormalities; first dose observation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride; Gelatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fingolimod (Experimental): Fingolimod 0.5 mg by mouth once daily for 7 days.
  Interventions: Drug: FTY720

INTERVENTIONS:
Drug: FTY720
  Other Names: 0.5 mg gelatin capsules

SUMMARY:
This study evaluated bradycardiac events during first dose observation of fingolimod in MS patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with relapsing remitting MS.
* Patients with highly active disease despite a full and adequate course of treatment with at least one disease modifying therapy.
* Patients who had been previously on 2nd line therapies. It was understood that these patients satisfied the above mentioned criteria listed under a. in the past.

This also included patients, who were previously treated with fingolimod (regardless of whether or not they had already been treated within the START study) but discontinued treatment due to medical reasons.

- or patients with rapidly evolving severe RRMS (e.g. > 2 relapses with disease progression in one year and > 1 Gd-enhancing lesion or with a significant increase in T2 lesions compared to a recent MRI).

Key Exclusion Criteria:

* immunocompromised patients
* active infections
* pregnant or nursing women, women of childbearing potential unless using 2 reliable forms of contraception
* presence of malignancy (other than localized basal cell carcinoma of the skin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6998 (Actual)
Dates: Start 2012-04-29 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (186):
- Germany (186):
  - Novartis Investigative Site, Ostfildern, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Altenholz-Stift, Germany
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Flensburg, Schleswig-Holstein
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Aalen
  - Novartis Investigative Site, Aalen-Wasseralfingen
  - Novartis Investigative Site, Abensberg
  - Novartis Investigative Site, Achim
  - Novartis Investigative Site, Aichach
  - Novartis Investigative Site, Altenburg
  - Novartis Investigative Site, Alzenau in Unterfranken
  - Novartis Investigative Site, Andernach
  - Novartis Investigative Site, Asbach
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Bad Hersfeld
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Honnef
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bad Wildbad
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berg
  - Novartis Investigative Site, Bergisch Gladbach
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bogen
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Borna
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Bruchsal
  - Novartis Investigative Site, Buchholz
  - Novartis Investigative Site, Buchholz in der Nordheide
  - Novartis Investigative Site, Butzbach
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Delbrück
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dillingen
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eberswalde
  - Novartis Investigative Site, Eisenach
  - Novartis Investigative Site, Eisleben Lutherstadt
  - Novartis Investigative Site, Eltville
  - Novartis Investigative Site, Emden
  - Novartis Investigative Site, Emmendingen
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Eschwege
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Gelnhausen
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Gilching
  - Novartis Investigative Site, Gladenbach
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Grevenbroich
  - Novartis Investigative Site, Griesheim
  - Novartis Investigative Site, Guelders
  - Novartis Investigative Site, Gummersbach
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Haar
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Halle S
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heidenheim
  - Novartis Investigative Site, Herdecke
  - Novartis Investigative Site, Herford
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Hoppegarten
  - Novartis Investigative Site, Ibbenbueren
  - Novartis Investigative Site, Idar-Oberstein
  - Novartis Investigative Site, Isselburg-Anholt
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Jülich
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Kaltenkirchen
  - Novartis Investigative Site, Kandel
  - Novartis Investigative Site, Karlstadt am Main
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Klingenmünster
  - Novartis Investigative Site, Koeln-Longerich
  - Novartis Investigative Site, Korbach
  - Novartis Investigative Site, Königsbrück
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Landshut
  - Novartis Investigative Site, Lappersdorf
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Lohr a. Main
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Lünen
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Meisenheim
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Mittweida
  - Novartis Investigative Site, Mosbach
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nagold
  - Novartis Investigative Site, Naumburg
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neuburg an der Donau
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Neusäß
  - Novartis Investigative Site, Neustadt an der Weinstraße
  - Novartis Investigative Site, Nordhausen
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Oldenburg I. Holstein
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Öhringen
  - Novartis Investigative Site, Paderborn
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Prien am Chiemsee
  - Novartis Investigative Site, Quakenbrück
  - Novartis Investigative Site, Querfurt
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Saint Ingbert
  - Novartis Investigative Site, Sande
  - Novartis Investigative Site, Schwalmstadt-Treysa
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Sinsheim
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Stralsund
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Telgte
  - Novartis Investigative Site, Teupitz
  - Novartis Investigative Site, Troisdorf
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Wasserburg
  - Novartis Investigative Site, Wendlingen
  - Novartis Investigative Site, Wermsdorf
  - Novartis Investigative Site, Westerstede
  - Novartis Investigative Site, Westerstede/Oldenburg
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wolfratshausen
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Würzburg
  - Novartis Investigative Site, Zwickau

REFERENCES:
- [Derived] Limmroth V, Ziemssen T, Lang M, Richter S, Wagner B, Haas J, Schmidt S, Gerbershagen K, Lassek C, Klotz L, Hoffmann O, Albert C, Schuh K, Baier-Ebert M, Wendt G, Schieb H, Hoyer S, Dechend R, Haverkamp W. Electrocardiographic assessments and cardiac events after fingolimod first dose - a comprehensive monitoring study. BMC Neurol. 2017 Jan 18;17(1):11. doi: 10.1186/s12883-016-0789-7. PMID 28100182

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6998 participants were enrolled into the study and were considered as part of the safety set, but 2 participants discontinued from the study and did not take any study drug.
Period: Overall Study
Arm/Group | Fingolimod
Started | 6998
Completed | 6961
Not Completed | 37
Not completed — Study completion was not documented. | 1
Not completed — Protocol deviation | 1
Not completed — Administrative problems | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4
Not completed — Abnormal test procedure results | 1
Not completed — Adverse Event | 24

BASELINE CHARACTERISTICS:
Arm/Group | Fingolimod
Number analyzed (Participants) | 6998
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4924
  Male | 2074

OUTCOME MEASURES:

1. Primary Outcome: Participants With 2nd or 3rd Degree Atrioventricular (AV) Block
Description: AV Blocks/Heart block is an abnormal heart rhythm where the heart beats too slowly; the electrical signals that tell the heart to contract are partially intermittent (Type 2:1) or slowed (1st and 2nd degree) or blocked (3rd degree) between the upper chambers (atria) and the lower chambers (ventricles). In 2nd degree AV Blocks, electrical impulses are intermittent (type 2:1) or delayed w/ each subsequent heartbeat (Mobitz type I) until a beat fails to reach the ventricles entirely. This type of block often is physiologic and observed in a highly relaxed state & during sleep. In 2nd degree AV Blocks type II, the atria electrical impulses are unable to reach the ventricles, a more serious condition. In 3rd degree AV Blocks (complete heart block), none of the electrical impulses reach either the atria or the ventricles. Patients can experience simultaneously both types of 2nd or 3rd degree AV Blocks without any symptoms.
Time Frame: baseline, during 6 hour monitoring post first dose observation
Population: Safety set: The safety set consisted of all enrolled participants for whom safety information was collected. Two patients of the safety analysis set discontinued the study without having received treatment, but safety information was collected on these two patients.
Measure: Number; unit: Participants
Arm/Group | Fingolimod
Number analyzed (Participants) | 6998
Participants
  Any AV block ll degree or higher | 120
  AV block ll degree: Mobitz type I degree | 117
  AV block II degree: Mobitz type II degree | 0
  AV block II degree: 2:1 | 43
  AV block III degree | 1

2. Primary Outcome: Number of Patients With Heart Rate Below 45 Beats Per Minute (BPM)
Description: Number of patients with heart rate below 45 beats bpm in ECG during first dose observation
Time Frame: baseline during 6 hour monitoring post dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Fingolimod
Number analyzed (Participants) | 6998
Participants | 63

3. Secondary Outcome: Number of Participants With Prolonged QTc Interval (Friderica)
Description: Number of patients with conduction abnormalities such as QT prolongation, first degree AV block during treatment initiation.
  The QT interval is a period between the activation and the regeneration of ventricular contraction. A prolonged QT interval can be a potential marker of cardiac arrhythmias.
  Two patients of the safety analysis set discontinued the study without having received treatment, but safety information was collected on these two patients.
Time Frame: baseline post-dose
Population: The safety set, which consisted of all enrolled participants for whom safety information was collected, was considered for the analysis. Only participants, who had baseline post-dose QTc interval data, were analyzed.
  Of the 6998 patients, 6844 patients had complete baseline post-dose QTc interval data.
Measure: Number; unit: Participants
Arm/Group | Fingolimod
Number analyzed (Participants) | 6844
Participants
  Female, QTcFridericia Interval > 470 ms: number analyzed (Participants) | 4808
  Female, QTcFridericia Interval > 470 ms | 7
  Male, QTcF Interval > 450 ms: number analyzed (Participants) | 2036
  Male, QTcF Interval > 450 ms | 6

4. Secondary Outcome: Number of Participants With Bradyarrhythmic Electrocardiogram (ECG) Events
Description: The number of participants with bradyarrhythmic electrocardiogram (ECG) events was assessed. Bradyarrhythmic ECG events are defined as QTc Fridericia time > 450 ms for males and > 470 ms for females.
Time Frame: up to day 7
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Fingolimod
Number analyzed (Participants) | 6998
Participants | 26

5. Secondary Outcome: Number of Patients With Cardiac Adverse Events
Description: The number of participants with the occurrence of subsequent cardiac adverse events (AEs) and serious cardiac AEs during study was assessed. Cardiac events were defined as the following Medical Dictionary for Regulatory Activities (MedDRA) preferred terms: angina pectoris, chest discomfort, dizziness, dyspnoea, dyspnoea exertional, fatigue, palpitations, syncope, vertigo, vertigo positional and vision blurred.
Time Frame: 7 days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Fingolimod
Number analyzed (Participants) | 6998
Participants
  Cardiac events | 489
  Serious cardiac AEs | 9

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for each patient from first administration of study drug until end of study visit, usually for one week. Furthermore, serious suspected adverse drug reactions (SADRs) had to be documented until 6 weeks after the patient has stopped study participation.
Arm/Group | Fingolimod
Serious Adverse Events (participants affected / at risk) | 160/6998
Other Adverse Events (participants affected / at risk) | 2179/6998
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=6998)
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Atrioventricular block complete (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 49
Bradycardia (Cardiac disorders) | 24
Coronary artery disease (Cardiac disorders) | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 2
Supraventricular extrasystoles (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Macular oedema (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
CD4/CD8 ratio decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 1
Heart rate decreased (Investigations) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Embolic cerebral infarction (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 26
Optic neuritis (Nervous system disorders) | 3
Partial seizures (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Subdural hygroma (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Borderline personality disorder (Psychiatric disorders) | 1
Depression suicidal (Psychiatric disorders) | 1
Mental fatigue (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Calculus urethral (Renal and urinary disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Blood pressure fluctuation (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=6998)
Anaemia (Blood and lymphatic system disorders) | 4
Eosinopenia (Blood and lymphatic system disorders) | 7
Eosinophilia (Blood and lymphatic system disorders) | 12
Granulocytosis (Blood and lymphatic system disorders) | 1
Haemoglobinaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 68
Lymphadenopathy (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 119
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Monocytopenia (Blood and lymphatic system disorders) | 4
Monocytosis (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 9
Neutrophilia (Blood and lymphatic system disorders) | 5
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Angina pectoris (Cardiac disorders) | 11
Arrhythmia (Cardiac disorders) | 7
Atrioventricular block first degree (Cardiac disorders) | 116
Atrioventricular block second degree (Cardiac disorders) | 74
Bradycardia (Cardiac disorders) | 48
Bundle branch block right (Cardiac disorders) | 1
Cardiac discomfort (Cardiac disorders) | 2
Cardiovascular disorder (Cardiac disorders) | 3
Coronary artery stenosis (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 4
Palpitations (Cardiac disorders) | 26
Pericardial effusion (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 8
Sinus tachycardia (Cardiac disorders) | 2
Supraventricular extrasystoles (Cardiac disorders) | 10
Tachycardia (Cardiac disorders) | 6
Ventricular extrasystoles (Cardiac disorders) | 4
Ventricular pre-excitation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 3
Ear pain (Ear and labyrinth disorders) | 3
External ear inflammation (Ear and labyrinth disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 68
Vertigo positional (Ear and labyrinth disorders) | 1
Amblyopia (Eye disorders) | 2
Blepharospasm (Eye disorders) | 1
Cataract (Eye disorders) | 1
Diplopia (Eye disorders) | 2
Eye irritation (Eye disorders) | 3
Eye pain (Eye disorders) | 11
Eye swelling (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 3
Foreign body sensation in eyes (Eye disorders) | 1
Iridocyclitis (Eye disorders) | 1
Macular oedema (Eye disorders) | 2
Ocular discomfort (Eye disorders) | 6
Photopsia (Eye disorders) | 1
Retinal vein thrombosis (Eye disorders) | 1
Vision blurred (Eye disorders) | 20
Visual acuity reduced (Eye disorders) | 3
Visual impairment (Eye disorders) | 6
Abdominal discomfort (Gastrointestinal disorders) | 9
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 53
Anal incontinence (Gastrointestinal disorders) | 2
Aphthous ulcer (Gastrointestinal disorders) | 1
Bowel movement irregularity (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 96
Dry mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 11
Dysphagia (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 9
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Gastrointestinal erosion (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 143
Odynophagia (Gastrointestinal disorders) | 1
Oral dysaesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Oral pruritus (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 2
Tongue blistering (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 13
Application site reaction (General disorders) | 1
Asthenia (General disorders) | 10
Chest discomfort (General disorders) | 24
Chest pain (General disorders) | 1
Chills (General disorders) | 11
Chronic fatigue syndrome (General disorders) | 3
Discomfort (General disorders) | 5
Face oedema (General disorders) | 2
Fatigue (General disorders) | 227
Feeling abnormal (General disorders) | 4
Feeling cold (General disorders) | 8
Feeling drunk (General disorders) | 1
Feeling hot (General disorders) | 5
Gait disturbance (General disorders) | 5
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 19
Infusion site inflammation (General disorders) | 1
Infusion site necrosis (General disorders) | 1
Local swelling (General disorders) | 1
Malaise (General disorders) | 11
Mucosal dryness (General disorders) | 1
Non-cardiac chest pain (General disorders) | 31
Oedema peripheral (General disorders) | 7
Pain (General disorders) | 2
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 17
Secretion discharge (General disorders) | 1
Sensation of foreign body (General disorders) | 1
Sense of oppression (General disorders) | 1
Temperature intolerance (General disorders) | 2
Thirst (General disorders) | 2
Hepatic steatosis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 5
Liver disorder (Hepatobiliary disorders) | 1
Food allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Seasonal allergy (Immune system disorders) | 1
Anal abscess (Infections and infestations) | 1
Anorectal infection (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 7
Chronic sinusitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 6
Dysentery (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 5
Genital herpes (Infections and infestations) | 1
Genitourinary tract infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 2
Helminthic infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 3
Herpes virus infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 4
Hordeolum (Infections and infestations) | 2
Infected bite (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 23
Laryngitis (Infections and infestations) | 3
Mastoiditis (Infections and infestations) | 1
Myelitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 137
Onychomycosis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 27
Pharyngitis (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 7
Rhinitis (Infections and infestations) | 12
Sialoadenitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 6
Tinea versicolour (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 15
Vaginal abscess (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Viral rhinitis (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 5
Animal bite (Injury, poisoning and procedural complications) | 1
Animal scratch (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Foot fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 21
Aspartate aminotransferase increased (Investigations) | 3
Basophil count increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 11
Blood chloride decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood glucose decreased (Investigations) | 2
Blood glucose increased (Investigations) | 9
Blood pressure decreased (Investigations) | 1
Blood pressure diastolic decreased (Investigations) | 3
Blood pressure diastolic increased (Investigations) | 2
Blood pressure increased (Investigations) | 10
Blood pressure systolic increased (Investigations) | 3
Blood urea increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Electrocardiogram P wave abnormal (Investigations) | 1
Electrocardiogram QRS complex prolonged (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 9
Electrocardiogram ST segment abnormal (Investigations) | 1
Electrocardiogram ST segment depression (Investigations) | 2
Electrocardiogram T wave inversion (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Eosinophil count decreased (Investigations) | 13
Eosinophil count increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 8
Haematocrit decreased (Investigations) | 1
Haematocrit increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 3
Haemoglobin increased (Investigations) | 1
Heart rate abnormal (Investigations) | 1
Heart rate decreased (Investigations) | 13
Heart rate increased (Investigations) | 7
Hepatic enzyme increased (Investigations) | 14
Liver function test increased (Investigations) | 3
Lymphocyte count abnormal (Investigations) | 2
Lymphocyte count decreased (Investigations) | 36
Lymphocyte count increased (Investigations) | 1
Monocyte count decreased (Investigations) | 3
Monocyte count increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 6
Neutrophil count increased (Investigations) | 7
Platelet aggregation (Investigations) | 1
Platelet count decreased (Investigations) | 1
Pulse abnormal (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Transaminases increased (Investigations) | 3
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 3
White blood cell count decreased (Investigations) | 18
White blood cell count increased (Investigations) | 5
White blood cells urine (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 9
Food craving (Metabolism and nutrition disorders) | 1
Gluten sensitivity (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 46
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 6
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 2
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 16
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 2
Carpal tunnel syndrome (Nervous system disorders) | 3
Disturbance in attention (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 126
Dizziness exertional (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 21
Epilepsy (Nervous system disorders) | 2
Facial spasm (Nervous system disorders) | 1
Head discomfort (Nervous system disorders) | 6
Headache (Nervous system disorders) | 316
Hemiparesis (Nervous system disorders) | 1
Hyperaesthesia (Nervous system disorders) | 1
Hypertonia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 14
Lhermitte's sign (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 17
Migraine with aura (Nervous system disorders) | 2
Monoparesis (Nervous system disorders) | 3
Multiple sclerosis (Nervous system disorders) | 3
Multiple sclerosis relapse (Nervous system disorders) | 70
Muscle spasticity (Nervous system disorders) | 6
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 4
Orthostatic intolerance (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 29
Peroneal nerve palsy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Psychogenic pseudosyncope (Nervous system disorders) | 1
Radial nerve compression (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 3
Sciatica (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 5
Syncope (Nervous system disorders) | 5
Tension headache (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 9
Trigeminal neuralgia (Nervous system disorders) | 3
Visual field defect (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Pregnancy of unknown location (Pregnancy, puerperium and perinatal conditions) | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Device defective (Product Issues) | 1
Adjustment disorder (Psychiatric disorders) | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 19
Dyssomnia (Psychiatric disorders) | 1
Emotional disorder (Psychiatric disorders) | 1
Initial insomnia (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 12
Irritability (Psychiatric disorders) | 2
Laziness (Psychiatric disorders) | 1
Listless (Psychiatric disorders) | 4
Mental disorder (Psychiatric disorders) | 1
Mental fatigue (Psychiatric disorders) | 2
Middle insomnia (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 3
Mood swings (Psychiatric disorders) | 2
Nervousness (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 7
Persistent depressive disorder (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 8
Sleep disorder (Psychiatric disorders) | 18
Bladder dysfunction (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 2
Nephritis (Renal and urinary disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Urge incontinence (Renal and urinary disorders) | 1
Breast discomfort (Reproductive system and breast disorders) | 2
Breast disorder (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Breast tenderness (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 3
Metrorrhagia (Reproductive system and breast disorders) | 1
Ovulation pain (Reproductive system and breast disorders) | 1
Priapism (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 2
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 15
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 4
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14
Night sweats (Skin and subcutaneous tissue disorders) | 3
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 24
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 15
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 2
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2
Walking disability (Social circumstances) | 1
Blood pressure fluctuation (Vascular disorders) | 2
Circulatory collapse (Vascular disorders) | 1
Diastolic hypertension (Vascular disorders) | 1
Flushing (Vascular disorders) | 4
Haematoma (Vascular disorders) | 1
Hot flush (Vascular disorders) | 3
Hypertension (Vascular disorders) | 64
Hypotension (Vascular disorders) | 12
Pallor (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 2
Varicose vein (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
292 centers were initiated but 278 centers randomized patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.